CLINICAL TRIAL: NCT01042002
Title: Effect of Exercise Before Gastric bypass-a Pilot Study
Brief Title: Effect of Exercise Before Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIT and gastric bypass
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Morbid Obesity
Keywords: High intensity exercise; morbid obesity; gastric bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity exercise (Experimental)
  Interventions: Behavioral: High intensity exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: High intensity exercise — High intensity exercise 3xweek for minimum 6 weeks
  Arms: High intensity exercise

SUMMARY:
Exercise training is proved to protect against premature cardiovascular mortality. Additionally there is evidence that relatively high exercise intensity may be an important factor for improving aerobic capacity and endothelial function in patients with post-infarction heart failure, metabolic syndrome, coronary artery disease, as well as in overweight and obese individuals.

The aims of this study is to investigate if High-intensity exercise before a gastric bypass operation will decrease hospitalization days and complications after the gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 20 years
* BMI: > 40 or > 35 with comorbidity
* Resident: Sør Trøndelag

Exclusion Criteria:

* Unstable Angina
* Resent cardiac infarction (within last year)
* heart failure
* Uncontrolled hypertension
* cardiomyopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hospitalization days after gastric bypass | Baseline, pre-operation and 6 months post operation

SECONDARY OUTCOMES:
Complications after gastric bypass | 6 months post operation

CONTACTS AND LOCATIONS:
Overall Officials: Arnt E Tjonna, PhD, Study Chair — Norwegain University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway